CLINICAL TRIAL: NCT06039007
Title: A run-in Study on the Safety and Tolerability of a Fasting Mimicking Diet in Relapsing Remitting Multiple Sclerosis (FAST-MS)
Brief Title: A run-in Study on the Safety and Tolerability of a Fasting Mimicking Diet in Relapsing Remitting Multiple Sclerosis
Acronym: FAST-MS
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAST-MS
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis
Keywords: fasting mimicking diet; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 7-DAY FMD (Experimental): The 7-DAY FMD by L-Nutra is a low-calorie and low-protein diet that provides all the necessary micronutrients to prevent malnutrition. This medically-designed dietary kit supplies food for 7 days, with Day 1 providing 1100 kcal, while days 2 to 5 provide 800 kcal per day. The diet consists of ingredients that are Generally Regarded As Safe (GRAS), selected for their fasting mimicking properties. Patients will take the 7-DAY FMD once every 60 days.
  Interventions: Dietary Supplement: 7-day Fasting-Mimicking Diet (7-DAY FMD)

INTERVENTIONS:
Dietary Supplement: 7-day Fasting-Mimicking Diet (7-DAY FMD) — This medically-designed dietary kit supplies food for 7 days, with Day 1 providing 1100 kcal, while days 2 to 5 provide 800 kcal per day.

SUMMARY:
This study is an open-label, single-arm, run-in study in patients with RRMS treated with first line therapies (interferon-beta, glatiramer acetate, teriflunomide and dimethyl fumarate), assessing the feasibility and tolerability of 3 cycles of Fasting-Mimicking Diet (FMD) over 6 months. All eligible patients will receive 3 cycles of the FMD once every 60 days in addition to their standard therapy with first line therapies. The diet provides 1100kcal on day 1 and 800 kcal on days 2-7. The diet consists of ingredients which are Generally Regarded As Safe (GRAS) selected for their fasting mimicking properties.

DETAILED DESCRIPTION:
The primary objective of the present study is to evaluate the safety and tolerability of 3 cycles of a 7 days FMD as a potential support to the management of patients affected by RRMS treated with first line therapies (interferon-beta, glatiramer acetate, teriflunomide and dimethyl fumarate). The primary endpoint is the number of serious and/or severe adverse events after the FMD start. A nutritionist will follow the patients for all the 6 months period, with the aim to monitor the FMD effects and to check for any possible problems. The nutritionist will call the patient on day 1 of every FMD cycle to answer any questions and check on the response, and on day 5 of the FMD to check on side effects and adherence.

At scheduled visits, vital signs and adverse events will be recorded from every patient.

Blood samples will be collected at baseline and just before at day 7 before returning to the normal diet on cycle 1 and 1 week after the first, the second and third FMD cycles. Should the patient display abnormal counts, the CBC will be repeated one week later. Additional FMD cycles will not be allowed in patients who do not return to normal levels of White Blood Cells (WBC) and Red Blood Cells (RBC).

At scheduled visits, vital signs and adverse events will be recorded from every patient.

FMD will be administered at month 0, month 2 and month 4 (3 cycles). MRI will be done at baseline and at month 6. At baseline and at month 6 patients will be evaluated with the EDSS and MSFC Functional composite scale. At the same time points, patients will be examined for the presence of cognitive disturbances by the Brief International Cognitive Assessment in Multiple Sclerosis (BICAMS) battery , of anxiety and depressive symptoms by the Hospital Anxiety and Depression Scale (HADS) , of fatigue by the Modified Fatigue Impact Scale (MFIS) , while quality of life will be monitored using the Short Form 36 Health Survey (SF-36) . A nutritional assessment will be carried out at enrollment and before every FMD cycle: patients will be examined evaluating the height and weight, with determination of the BMI; the bodily composition will be measured with a dynamometer and by BIA.

Adverse events (AEs) will be monitored for each patient up to the study termination; in case of ongoing AEs at study end, patients will be followed for 30 additional days.

During the whole duration of the study, patients will be instructed to perform standardized physical exercises, in order to avoid fasting induced sarcopenia. Briefly, before each FMD cycle, patients will be recommended to exercise 30 minutes daily according to a dedicated training program to improve their muscle anabolism in the interval between the three FMD cycles.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RRMS (Thompson et al. 2018);
* Disease duration 6 months to 10 years (included);
* EDSS 0 to 4, 5;
* Treatment with first line therapies (interferon-beta, glatiramer acetate, teriflunomide and dimethyl fumarate).

Exclusion Criteria:

* < 6 months since treatment start with first line therapies (interferon-beta, glatiramer acetate, teriflunomide and dimethyl fumarate);
* Relapse < 60 days;
* Any active or chronic infection;
* Previous history of a malignancy other than basal cell carcinoma of the skin or carcinoma in situ that has been in remission for more than one year;
* Severely limited life expectancy by another co-morbid illness;
* Nutritional risk screening (NRS 2002) > or = 3;
* BMI <= 18.5 kg/m2;
* Bio-impedance phase angle <5.0°;
* History of previous diagnosis of myelodysplasia or previous hematologic disease or current clinically relevant abnormalities of white blood cell counts;

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of 7-day FMD | 6 months
  Safety of 7-day FMD in terms of percentage of patients experiencing adverse events and/or worsening of nutritional status.
  To obtain clinical data on safety of the FMD in MCI or AD patients as assessed by percentage of patients (%) experiencing > grade 3 adverse events and/or a significant decrease in their lean body mass (kg) and/or with a reduction of phase angle <5° assessed with bio-impedance measurements. for Adverse Events (CTCAE)

SECONDARY OUTCOMES:
Percentage of patients able to achieve the designated diet regimen | 6 months
  Feasibility of FMD in terms of percentage of patients able to complete the diet regimen To evaluate the feasibility of the FMD in MCI and AD patients as assessed by the percentage of patients (%) able to achieve the designated diet regimen.
Changes in the Expanded Disability Status Scale (EDSS) | 6 months
  Score 0-10
Changes in Body Mass Index (BMI) | 6 months
  kg/m2
Changes in the serum light chain neurofilaments concentration | 6 months
  ng/ml
White Blood Cells | 6 months
  mil/mm3
Efficacy of the FMD in terms of nutritional state | 6 months
  Efficacy of the FMD in terms of nutritional state will be assessed with phase angle with bioimpedance (°)

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Martino, Genova, Italy